CLINICAL TRIAL: NCT04460027
Title: Woebot for Substance Use Disorders During COVID-19
Brief Title: W-SUDs for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Woebot Health (Industry)
Collaborators: Stanford University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56439; 4R44DA048712-02 (NIH)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Substance Use Disorders; Alcohol Use Disorder
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-SUDs (Experimental)
  Interventions: Other: Woebot Substance Use Disorder
- Wait List Control (No Intervention)

INTERVENTIONS:
Other: Woebot Substance Use Disorder — Woebot Substance Use Disorder is an automated conversational agent, available through a smartphone application, that delivers evidence-based psychotherapeutics, empathy, and emotional health psychoeducation.
  Arms: W-SUDs

SUMMARY:
The purpose of this study is to test the efficacy of a substance use disorder intervention delivered via a mobile application in an adult population during the COVID-19 pandemic.

This study that will test the comparative efficacy of the mobile-app based substance use disorder program to reduce substance use relative to a wait list control condition, and explore between group differences on quality of life indices as well as retention and engagement during COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* All genders aged 18-65 years
* Access to a smartphone
* Available and committed to engage with app and complete assessments
* Be willing to provide email address (as this is how assessment incentives will be distributed),
* Literate in English (as W-SUDs conversational and video materials will be in English).

Exclusion Criteria:

* Pregnancy (as W-SUDs will not be specifically developed to address the unique needs of this population)
* History of severe drug/alcohol use
* History of opioid misuse without medication-assisted treatment
* Suicide attempt within the past year
* Opioid overdose within the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Waitlist Control: Participants randomized to the waitlist control arm were provided access to W-SUDs after completing the 8-week study.
Period: Overall Study
Arm/Group | W-SUDs | Waitlist Control
Started | 88 | 92
Completed | 71 | 81
Not Completed | 17 | 11

BASELINE CHARACTERISTICS:
Groups:
- Wait List Control: Participants randomized to the waitlist control arm were provided access to W-SUDs after completing the 8-week study.
- Total: Total of all reporting groups
Arm/Group | W-SUDs | Wait List Control | Total
Number analyzed (Participants) | 88 | 92 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (12.1) | 39.8 (11.2) | 40.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 30 | 33 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 76 | 80 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 70 | 70 | 140
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Substance Use Occasions in the Past 30 Days From Baseline to Post-treatment at 8 Weeks
Description: Change in number of substance use occasions in the past 30 days from Baseline to Post-treatment at 8 weeks
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: occasions
Arm/Group | W-SUDs | Waitlist Control
Number analyzed (Participants) | 71 | 81
occasions | -9.1 (2.0) | -4.7 (1.0)

2. Secondary Outcome: Change in Short Inventory of Problems - Alcohol and Drugs (SIP-AD) From Baseline to Post-treatment at 8 Weeks
Description: Measure of substance use problems. The SIP-AD assesses substance use problems in the past 30 days. Total score consists of of the sum of all 15 items, ranging from 0-45, where greater scores indicate greater substance use problems.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
score on a scale | -5.3 (1.1) | -4.7 (1.0)

3. Secondary Outcome: Change in Drug Abuse Screening Test (DAST-10) From Baseline to Post-treatment at 8 Weeks
Description: Measure of drug abuse related consequences. The DAST-10 is a brief, 10-item self-report measure that assesses consequences related to drug abuse, excluding alcohol and tobacco. The range is 0-10, where higher scores indicate greater severity. Adapted from past 12 months to past 30 days.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
score on a scale | 1.3 (1.8) | 2.2 (2.1)

4. Secondary Outcome: Change in Brief Situational Confidence Questionnaire (BSCQ) From Baseline to Post-treatment at 8 Weeks
Description: Measure of self-confidence. The 8-item BSCQ is a state dependent measure that assesses self-confidence to resist the urge to drink heavily or use drugs in a variety of situations. Each of the 8 scale situations consists of a 100-mm line, anchored by 0% ("not at all confident") and 100% ("totally confident") where clients are asked to indicate confidence on a scale from 0% to 100%. Higher scores are associated with greater confidence.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
score on a scale | 11.8 (3.4) | 5.3 (3.1)

5. Secondary Outcome: Change in Craving Ratings From Baseline to Post-treatment at 8 Weeks
Description: A one-item, self-reported rating of craving intensity to use substances over the past 7 days. Score ranges is from 0-4, where a greater score indicates a more intense urge to use.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
scores on a scale | -.5 (.1) | -.4 (.1)

6. Secondary Outcome: Change in Pain Ratings From Baseline to Post-treatment at 8 Weeks
Description: A one item, self-reported rating of pain. Scores range from 0-100 where higher scores indicate greater levels of pain.
Time Frame: Change from Baseline to Post-treatment at 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
units on a scale | -5.1 (2.8) | -.8 (2.5)

7. Secondary Outcome: Change in Patient Health Questionnaire-8 (PHQ-8) From Baseline to Post-treatment at 8 Weeks
Description: Measure of depression. An 8-item self-report questionnaire that assesses the frequency and severity of depression symptoms. Total scores range from 0 to 24 where higher scores indicate greater levels of depression.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
units on a scale | -1.6 (.6) | -1.7 (.6)

8. Secondary Outcome: Change in General Anxiety Disorder (GAD-7) From Baseline to Post-treatment at 8 Weeks
Description: Measure of anxiety. A 7-item brief self-report measure used to assess the frequency and severity of anxious thoughts and behaviors over the past 2 weeks. Total score between 0-21, where higher scores indicate greater levels of anxiety.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
units on a scale | -1.6 (.6) | -.7 (.5)

9. Secondary Outcome: Change in CAIR Pandemic Impact Questionnaire (CAIR-PIQ) From Baseline to Post-treatment at 8 Weeks
Description: Assesses impact of the COVID-19 pandemic in terms of exposure to stressors, mental health impact, and growth. Possible total score range from 0-22, where greater scores are related to greater impact.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | W-SUDs | Wait List Control
Number analyzed (Participants) | 71 | 81
units on a scale | -1.8 (.5) | -1.4 (.5)

10. Secondary Outcome: Client Satisfaction Questionnaire (CSQ) at Post-treatment at 8 Weeks
Description: Measure of satisfaction. An 8-item measure used to assess client's satisfaction with treatment on a 4-point scale. Example questions include, "How would you rate the quality of service you received"? and "Did you get the kind of service you wanted?" Total sums range from 8-32, with high scores indicating greater satisfaction with the W-SUDs mobile application.
Time Frame: Post-treatment (8 weeks from Baseline)
Population: This measure was administered to the active intervention arm only; assessment not applicable for a waitlist control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs
Number analyzed (Participants) | 71
score on a scale | 25.5 (5.0)

11. Secondary Outcome: Usage Rating Profile - Intervention (URPI)-Acceptability at Post-treatment at 8 Weeks
Description: Measure of acceptability. A 6-item subscale that inquires about intervention acceptability. Total scores range from 6-36, where greater scores indicate greater intervention acceptability.
Time Frame: Post-treatment (8 weeks from Baseline)
Population: This measure was administered to the active intervention arm only; assessment not applicable for a waitlist control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs
Number analyzed (Participants) | 71
score on a scale | 29.0 (4.8)

12. Secondary Outcome: Usage Rating Profile - Intervention (URPI)-Feasibility at Post-treatment at 8 Weeks
Description: Measure of feasibility. A 6-item subscale that inquires about factors that impact treatment usage (i.e., intervention quality). Total scores range from 6-36, where greater scores indicate greater intervention feasibility.
Time Frame: Post-treatment (8 weeks from Baseline)
Population: This measure was administered to the active intervention arm only; assessment not applicable for a waitlist control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs
Number analyzed (Participants) | 71
score on a scale | 32.0 (3.6)

13. Secondary Outcome: Change in Working Alliance Inventory (WAI-SR) From Mid-treatment at 4 Weeks to Post-treatment at 8 Weeks
Description: Measure of working alliance. A measure of therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Total scores range from 12-60, with higher scores indicating greater alliance. The present study utilized the validated 12-item Short-Revised version (WAI-SR) with minor changes to language, replacing "therapist" with "Woebot".
Time Frame: Change from Mid-treatment at 4 weeks to Post-treatment at 8 weeks
Population: This measure was administered to the active intervention arm only; assessment not applicable for a waitlist control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs
Number analyzed (Participants) | 71
score on a scale | 44.0 (12.5)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed at post-treatment, 8 weeks from baseline.
Description: Serious adverse events occurring during treatment were assessed for hospitalization related to substance use, suicide attempt, alcohol or drug overdose, and severe withdrawal (eg, delirium tremens). Positive endorsements were followed up with questions about the timing, diagnosis, and resolution. If additional details were needed to determine whether the event was study related, a team member reached out to the participant.
Arm/Group | W-SUDs | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/88 | 1/92
Other Adverse Events (participants affected / at risk) | 0/88 | 0/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | W-SUDs (N=88) | Wait List Control (N=92)
Hospitalization (General disorders) | 0 (0) | 1 (1) — Hospitalization for alcohol detoxification

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT04460027/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04460027/SAP_001.pdf
  • Informed Consent Form (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT04460027/ICF_002.pdf